CLINICAL TRIAL: NCT01305382
Title: Noninvasive Evaluation of Cardiac Allograft Vasculopathy in Heart Transplant Recipients II
Brief Title: Noninvasive Evaluation of Cardiac Allograft Vasculopathy
Acronym: CAVII
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0808M43361
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Cardiac Allograft Vasculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Heart Transplant Cohort: This group consist of transplant subjects within 10 years of heart transplant
- Heart Failure Sub group: Consist of subjects with advanced heart failure (NYHA class III and IV)
- Healthy Volunteer: This groups consist of healthy individuals

SUMMARY:
Abnormal peripheral endothelial function and alterations in circulating biomarkers that are associated with endothelial activation and inflammation correlate with angiographic evidence of cardiac allograft vasculopathy, defined as greater than 25% stenosis in a major coronary artery.

DETAILED DESCRIPTION:
Cardiac transplantation has become the established treatment of choice for eligible patients with end-stage heart failure. Cardiac allograft vasculopathy (CAV) is a major and potentially preventable limitation to long-term survival in cardiac transplant recipients. CAV affects up to 50% of recipients by year 5, though intimal thickening is present in up to 58% one year after transplantation. CAV is characterized by diffuse, concentric intimal hyperplasia, involving both epicardial and intramyocardial coronary arteries. In its most advanced stages, CAV is not amenable to standard revascularization procedures making the only cure re-transplantation. Given the limited donor pool and poor outcome, re-transplantation is not an option for all patients. CAV tends to be a silent process. Due to denervation of the transplanted heart, transplant recipients do not typically have chest pain, and thus the first symptoms of CAV may be those of heart failure or sudden cardiac death. Traditional risk factors are important in predicting the development of CAV, however non-traditional risk factors appear equally important and include cellular and humoral rejection, graft ischemia at the time of implantation, and cytomegalovirus (CMV).

Despite the specific inciting event, the end result is endothelial dysfunction, which is the predecessor to CAV. Methods to detect, prevent, and treat endothelial dysfunction and subsequently CAV are few. The rapidity with which it develops, however, affords a great opportunity to study mechanisms and potential interventions in a relatively short period of time.

Chronic inflammation and immune activation and subsequent endothelial injury are felt to immunopathogenic in the development of CAV. Endothelial activation is a precursor to the development of transplant vasculopathy, and multiple biomarkers have been shown to correlate with the presence of endothelial dysfunction in transplant vasculopathy. (fig. 1) Endothelial activation, as determined by the presence of adhesion molecules, begins hours after brain death in a donor. VCAM-1, e-selectin, and p-selectin are expressed early after brain death in the donor and are elevated throughout transplantation in the recipient as a response to injury in the donor heart. P-selectin and VCAM remain elevated while e-selectin gradually decrease over three months. There is data suggesting that p-selectin and VCAM remain elevated up to 2 years after transplantation, suggesting persistent inflammation and immune activation after transplant. Furthermore, nitric oxide is the principal mediator of protective effects on the endothelium. The nitric oxide pathway is essential in maintaining vascular integrity in cardiac recipients, and inhibition of this pathway accelerates intimal thickening and worsens endothelial function caused by rejection. Intimal thickening is a marker of endothelial dysfunction and a precursor to the development of CAV.

Thus, these markers and others involved in atherogenesis, remodeling, immune activation and endothelial activation, may provide a useful modality in predicting the presence of vasculopathy. In addition, studying various components of the process, eg. inflammation and injury, will provide much needed information regarding targets for therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Provide informed consent
* Presence of advanced heart failure (NYHA class III, IV) on medical therapy
* Patients with advanced heart failure on transplant list
* Transplant recipients undergoing invasive evaluation for coronary artery disease within 6 months to ten years post transplantation

Exclusion Criteria:

* Current tobacco use
* History of chronic kidney disease
* Active infection
* History of organ transplantation
* Diabetes Mellitus
* History of Hypertension
* Known coronary artery disease
* Connective tissue disorder
* History of hyperlipidemia
* History of Migraine or Chronic unevaluated headaches
* Patients with chronic kidney disease stage 4 defined as GFR<30 mL/min/1.73 m2 or acute renal failure
* Patients with acute rejection, Grade 3A or greater
* Active infection
* Re-transplant or Multi-organ transplant recipient
* Surgery within 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart Transplant subjects within 10 years of heart transplantation Subjects with advanced heart failure Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Stenosis of a major coronary artery greater than 25% on coronary angiogram. | 1 year
  The purpose of this study is to determine whether certain levels and patterns of expression of biomarkers known to be related to endothelial function and abnormalities in peripheral artery function are predictive of the presence of transplant vasculopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Monica M Colvin-Adams, MD, MS, Principal Investigator — Cardiology, University of Minnesota
Locations (1):
- Cardiology Division, University of Minnesota, Minneapolis, Minnesota, United States